CLINICAL TRIAL: NCT01712022
Title: Evaluation of Corneal Epithelial Thickness Mapping
Status: Completed | Type: Observational
Sponsor: Optovue (Industry)
Responsible Party: Sponsor
Other Study IDs: 200-48071
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Dry Eye and Contact Lens Wear
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Dry Eye: clinical diagnosis of dry eye
- Contact Lens: routine wear of contact lens
- Normal: Not having history of dry eye or contact lens wear or corneal pathology or surgery

SUMMARY:
Optovue has developed a new feature for mapping corneal epithelial thickness. The purpose of the study is to evaluate the accuracy and repeatability of the epithelial thickness measurement. Consented subjects will undergo a series of cornea measurements using optical coherence tomography (OCT) that will be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able and willing to provide consent
* Able and willing to complete the required examinations
* DRY EYE GROUP ONLY: Clinical diagnosis of dry eye
* CONTACT LENS GROUP ONLY: Regular contact lens wear

Exclusion Criteria:

* History of ocular surgery
* History of laser refractive surgery
* History of cataract surgery
* DRY EYE GROUP ONLY: Corneal pathology not associated with dry eye
* CONTACT LENS GROUP ONLY: Corneal pathology including dry eye
* NORMAL GROUP ONLY: History of contact lens wear or dry eye or corneal pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: seeing eye doctor for routine or follow-up care
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
corneal epithelial thickness | Day 1

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Fishman Vision, Palo Alto, California
  - Gordon-Weiss-Schanzlin Vision Institute, San Diego, California
  - Brass Eye Center, Latham, New York